CLINICAL TRIAL: NCT01384565
Title: A Prospective Randomized Double Blind Trial to Study the Efficacy of G-CSF and Erythropoetin in Survival of Patients With Decompensated Liver Disease
Brief Title: G-CSF and Erythropoetin in Survival of Patients With Decompensated Liver Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILBS DLD 01
Record Dates: First submitted 2011-06-28; First posted 2011-06-29 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Chronic Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- G-CSF+EPO (Active Comparator)
  Interventions: Drug: G-CSF+EPO
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: G-CSF+EPO — Drug: Granulocyte Colony-stimulating Factor (G-CSF) and Erythropoetin (EPO)
  G-CSF (in prefilled syringe) at a dose of 5 µg/kg s/c at days 1, 2, 3, 4, 5 and then every 3rd day till day 28 (total 12 doses), along with Darbopoetin alpha 100 mcg/ week (in prefilled syringe) for 4 weeks (total 4 doses).
  Arms: G-CSF+EPO Drug: Placebo
  Placebo 1 (in prefilled syringe) s/c at days 1, 2, 3, 4, 5 and then every 3rd day till day 28 (total 12 doses), along with Placebo 2 every week (in prefilled syringe) for 4 weeks (total 4 doses).
  Arms: G-CSF+EPO
Drug: Placebo — Placebo 1 (in prefilled syringe) s/c at days 1, 2, 3, 4, 5 and then every 3rd day till day 28 (total 12 doses), along with Placebo 2 every week (in prefilled syringe) for 4 weeks (total 4 doses).
  Arms: Placebo

SUMMARY:
Study Design

50 patients will be enrolled and randomized into patients (Group IA) and controls (Group I B)

Investigations:

Hematology CBC, Prothrombin time and INR Peripheral smear, Retics Biochemistry Liver function testing, AFP Kidney function testing Etiology of chronic liver disease Infectious etiology: total antiHBc, anti HCV, HCV RNA, HBV DNA Non infectious etiology: Autoimmune markers, copper studies, iron studies, HOMA IR, FBS Etiology of decompensation Variceal bleed Infection ( blood culture, urine culture, sputum culture, chest xray) Surgery Drugs Alcohol intake Ascitic fluid analysis UGI endoscopy Imaging USG abdomen with Doppler for spleno-portal axis CECT- Triple phase upper abdomen Liver regenerative potential efficacy testing Histology ( by transjugular liver biopsy) Liver Dendritic cells ( CD11c, CD40, CD 54, CD 123, BDCA 2 staining) by flow cytometry CD 34+ cells, CD 45+ cells and CD 133+ cells measurement in hepatic venous blood, peripheral blood and liver biopsy by flow cytometry Markers of proliferation like Ki- 67, proliferating cell nuclear antigen (PCNA) in liver biopsy Markers of angiogenesis like VEGF, v WF in hepatic venous blood Measurement of Hepatic venous pressure gradient ( HVPG)

ELIGIBILITY:
Inclusion Criteria:

* All patients who were known to have cirrhosis of liver with portal hypertension, now decompensated with ascites/ jaundice/ bleed/ HE/ HRS

Exclusion Criteria:

* Age <12 or > 75 years

  * Autoimmune disorders
  * HCC
  * Sepsis ( Any culture positive: blood, urine, any other obvious source of infection: UTI, SBP)
  * Multi organ failure
  * Grade 4 HE
  * HIV seropositivity / pregnancy
  * Essential Hypertension
  * Patients being taken up for transplant
  * Refusal to participate in the study

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2011-07; Primary Completion 2012-11 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
transplant free survival at 1 year | 3 Months

SECONDARY OUTCOMES:
transplant free survival at 6 months, histo-pathological evidence of hepatic regeneration and mobilization of CD34/stem cells, improvement in severity assessment indices | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Shiv Kumar Sarin, MD,DM, Study Director — Institute of Liver & Biliary Sciences (ILBS)
Locations (1):
- Institute of liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Kedarisetty CK, Anand L, Bhardwaj A, Bhadoria AS, Kumar G, Vyas AK, David P, Trehanpati N, Rastogi A, Bihari C, Maiwall R, Garg HK, Vashishtha C, Kumar M, Bhatia V, Sarin SK. Combination of granulocyte colony-stimulating factor and erythropoietin improves outcomes of patients with decompensated cirrhosis. Gastroenterology. 2015 Jun;148(7):1362-70.e7. doi: 10.1053/j.gastro.2015.02.054. Epub 2015 Mar 4. PMID 25749502